CLINICAL TRIAL: NCT06834724
Title: Clinical Outcomes of Continuous Positive Airway Pressure Treatment in People With Obstructive Sleep Apnea
Brief Title: Clinical Outcomes of Continuous Positive Airway Pressure Treatment in People With Obstructive Sleep Apnea and Chronic Pain
Status: Recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Olivier Mairesse, Professor, Vrije Universiteit Brussel
Other Study IDs: 1
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Obstructive Sleep Apnea
Keywords: Chronic pain; Obstructive sleep apnoea; Obstructive sleep apnea; CPAP
MeSH Terms: conditions — Chronic Pain; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CPAP group: People defined as obstructive sleep apnoea with or without chronic pain. They undergo standard care (CPAP therapy).
  Interventions: Other: Standard OSA care

INTERVENTIONS:
Other: Standard OSA care — All people will undergo standard care.

SUMMARY:
The bidirectional link between sleep and pain is a widely accepted concept. While there has been much focus on this in recent years, studies investigating obstructive sleep apnoea (OSA) and chronic pain are still not very common, especially in context of continuous positive airway pressure (CPAP) therapy.

In this study, people recently diagnosed with OSA, a common sleep disorder, that are receiving a CPAP mask are asked to fill in questionnaires at baseline, 3- and 6-month follow-up. Data of people with and without chronic pain will be collected and we will use the data will allow us to answer a number of clinically relevant questions. The primary questions investigate the following: 1) The association of CPAP adherence and pain outcomes with CPAP therapy at 3-month follow-up; 2) The association of baseline Apnoea-Hyopnea-Index on pain outcomes with CPAP therapy at 3-month follow-up. Secondary questions investigate the relevance of co-morbid insomnia (COMISA), the influence of chronic pain on CPAP adherence and general clinical outcomes of CPAP therapy in people with chronic pain.

DETAILED DESCRIPTION:
In this study, participants with obstructive sleep apnoea (OSA) that start continuous positive airway pressure (CPAP) treatment will be asked to fill in questionnaires at baseline and two follow-up time points (3 and 6 months after the start of CPAP treatment). This information, information on CPAP adherence and information from the polysomnography assessment every participant has undergone prior to starting CPAP will allow us to investigate relevant outcomes of CPAP therapy in people with chronic pain. The detailed research questions are the following:

Primary research questions Longitudinal

1. Are average hours of CPAP use per night (continuous variable) associated with average pain intensity at 3-month follow-up in people with CP and OSA?
2. Is AHI at baseline associated with average pain intensity at 3-month follow-up in people with CP and OSA?

Secondary research questions Cross-sectional

1. Is there a difference in CPAP use in hours (measured at 3-month follow-up) between people with OSA-only, OSA and CP, OSA and comorbid insomnia (COMISA - defined via the Insomnia Severity Index ≥15) and COMISA with CP?
2. What is the prevalence of CP in patients with clinically relevant OSA in a sleep clinic setting?
3. Is there a difference in average pain intensity between people with OSA and CP and people with COMISA and CP?

Longitudinal

1. What are the short- (3 months) and long-term (6 months) clinical outcomes (average pain intensity, fatigue, sleepiness, sleep quality, depression, anxiety, quality of life) of CPAP treatment for patients with clinically relevant OSA and comorbid CP?
2. Does average pain intensity measured at 3 and 6-month follow-up differ between patients that show CPAP adherence (= use of CPAP for a minimum of four hours each night on at least 70% of the monitored nights) compared to patients with non-adherence (= use of CPAP for a less than four hours each night on at least 70% of the monitored nights)?
3. Is average pain intensity at baseline a predictor for CPAP adherence in people with CP and comorbid clinically relevant OSA as measured at 3-month follow-up.
4. Is there a difference in pain outcomes measured at follow-up points at 3 and 6 months between people with CP and COMISA compared to patients with only OSA and CP?
5. Is there a difference in self-reported health status with CPAP therapy at 3 and 6-month follow-up between people with clinically relevant OSA and CP compared to those without CP?
6. Are average hours of CPAP use per night (continuous variable) associated with average pain intensity at 6-month follow-up in people with CP and OSA?
7. Is AHI at baseline associated with average pain intensity at 6-month follow-up in people with CP and OSA?

Sensitivity and subgroup analyses will analyse data for people with headaches and other chronic pain separately considering headaches to be a very common direct consequence of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must be able to read and write in Dutch, French or English
* Participants must be diagnosed with clinically relevant OSA and newly start CPAP treatment:
* AHI ≥ 15
* Prescribed CPAP for the first time as a treatment for their OSA
* Participants must have read and signed the ICF

Exclusion Criteria:

* Participants who are currently receiving CPAP treatment or have had a CPAP treatment in the last year
* Participant receiving CPAP for other conditions than OSA (e.g. Central Sleep Apnoea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target group for the study consists of adult, Dutch, French or Englisch speaking patients who have been referred to the sleep clinic. These patients have been diagnosed with OSA and will start to receive CPAP treatment. They are included independent of their chronic pain status but some analyses will be done in sub-groups.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Average Pain during last 1 week | 3-months after initiation of CPAP therapy
  Participants are asked for the average pain they had during the last 1 week. They answer on a scale for 0-10 with 0 being no pain and 10 being the worst pain ever. This is a single question taken from the Brief Pain Inventory

SECONDARY OUTCOMES:
CPAP adherence | 3-months after initiation of CPAP therapy
  Average CPAP use in hours per night as measured by the CPAP device
Prevalence of chronic pain in people with OSA undergoing CPAP treatment | Baseline
  Chronic pain defined as pain anywhere in the body that is present every day or most days for 3 months or longer and that regularly impairs quality of life or ability to do activities (leisure, work).
Average Pain during last 1 week | 6-months after initiation of CPAP therapy
  Participants are asked for the average pain they had during the last 1 week. They answer on a scale for 0-10 with 0 being no pain and 10 being the worst pain ever. This is a single question taken from the Brief Pain Inventory
Fatigue (Mental and Physical) | 3 and 6 months after initiation of CPAP therapy
  Measured using the Brugmann Fatigue scale - 0-12 for each subscale (Mental fatigue and physical fatigue with 0 indicating no fatigue and 12 severe fatigue)
Sleepiness | 3 and 6 months after initiation of CPAP therapy
  Measured using the Epworth sleepiness scale - 0-24 with 0 indicating no sleepiness and 24 severe sleepiness.
Subjective sleep quality | 3 and 6 months after initiation of CPAP therapy
  Measured using the Pittsburgh Sleep quality index total score (0-21 with 0 indicating good sleep quality and 21 very bad sleep quality)
Depression | 3 and 6 months after initiation of CPAP therapy
  Measured using the depression subscale of the Hospital Anxiety and Depression Scale - 0-21 with 0 being no depressive symptomatology and 21 being severe depressive symptomatology
Anxiety | 3 and 6 months after initiation of CPAP therapy
  Measured using the anxiety subscale of the Hospital Anxiety and Depression Scale - 0-21 with 0 being no anxiety and 21 being severe anxiety
Self-reported health status | 3 and 6 months after initiation of CPAP therapy
  Measured using the Short Form 36 (SF-36) subscales with 0 indicating worse status and 100 indicating better health status in a domain

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No